CLINICAL TRIAL: NCT00011531
Title: Investigation of Subatmospheric Pressure Dressing on Pressure Ulcer Healing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Longaker, Michael - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2108R
Record Dates: First submitted 2001-02-22; First posted 2001-02-26 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2001-01

CONDITIONS: Diabetic Foot Ulcers
Keywords: Decubitus Ulcers; dehiscence; SCI; wound healing
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Prevention of Pressure Ulcers

INTERVENTIONS:
Procedure: Prevention of Pressure Ulcers

SUMMARY:
Many spinal cord injury (SCI) and otherwise debilitated patients develop pressure ulcers over the course of their injury or disease. Despite enhanced wound care management, many pressure ulcers do not heal completely and require surgical myocutaneous rotational flap coverage. Even then they often recur.

The objectives of this study are: (1) to conduct a controlled comparative study of the effectiveness of subatmospheric pressure dressing (SPD) in healing pressure ulcers versus conventional saline wet-to-moist dressing techniques; (2) to establish indications and contra-indications for use of SPD In treating pressure ulcers; and (3) to develop a noninvasive, clinically usable optical digitizer and associated software for measurement of wound geometry for standardized quantitative assessment and longitudinal monitoring of wound healing.

DETAILED DESCRIPTION:
Many spinal cord injury (SCI) and otherwise debilitated patients develop pressure ulcers over the course of their injury or disease. Despite enhanced wound care management, many pressure ulcers do not heal completely and require surgical myocutaneous rotational flap coverage. Even then they often recur.

HYPOTHESIS: Subatmospheric pressure dressing (SPD) treatment applied to pressure ulcers will either completely close them, or heal to a point allowing for skin graft coverage, more often than 0.9% normal saline wet-to-moist dressing (WTMD) treatment.

OBJECTIVES: The objectives of this study are: (1) to conduct a controlled comparative study of the effectiveness of subatmospheric pressure dressing (SPD) in healing pressure ulcers versus conventional saline wet-to-moist dressing techniques; (2) to establish indications and contra-indications for use of SPD In treating pressure ulcers; and (3) to develop a noninvasive, clinically usable optical digitizer and associated software for measurement of wound geometry for standardized quantitative assessment and longitudinal monitoring of wound healing.

RESEARCH METHODS: 120 patients with stage III or IV pressure ulcers meeting the project selection criteria will be recruited for the project. Patients will be randomly assigned in a 3:1 (SPD to WTMD) ratio to either the control group receiving 0.9% normal saline wet-to-moist wound dressing and treatment, or to the subatmospheric pressure dressing group. All subjects selected will be further stratified according to degree of wound severity, nutritional status, and evidence of wound infection. The WTMD group will receive 0.9% NS moistened gauze applied to the wound, which will be changed every 8 hours. The SPD group will receive SPD dressing with the VACTM system set at a constant subatmospheric pressure of negative 125 mmHg. The SPD device and dressing will be left in place and changed every Monday, Wednesday, and Friday. The subjects' pressure ulcers will be measured on day 0 and then on a weekly basis. Ulcer surface shape, area, and coloration will be recorded with a digital camera and also by tracing the ulcer perimeter on a flexible translucent plastic film with grid overlaid on the wound. In addition, an optical laser scanner will used to record ulcer shape, area, and coloration, and body/limb segmental volume in the region of the wound. Volume will also be measured using alginate wound impressions to form RTV silicone molds for fluid displacement measurement. The molds of the wounds will also be optically digitized and wound perimeter, topical surface area, total 3-D surface area, and volume calculated using computer image processing, planimetry, and volumetry software developed in the project. Local body/limb segment volume will also be calculated to monitor edematous fluctuations. Based on these measurements, the wound responses will be scored as described in Table 2 after one month or at the time of the patient's withdrawal from the study. The association between response level and treatment type will be analyzed using Chi-square test of association. Mantel-Haenszel Chi-square and logistic regression will be used to control for prognostic variables.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Wounds and ulcers

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2000-01; Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Longaker, MD, Principal Investigator — New York Harbor HCS
Locations (1):
- New York Harbor HCS, New York, New York, United States